CLINICAL TRIAL: NCT04639778
Title: Evaluation of a Personalized Care Path After Bariatric Surgery Based on Monitoring the Weight Evolution Using a Connected Scale
Brief Title: Monitoring the Weight Evolution Using a Connected Scale
Acronym: TELEBARIA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2017_78; 2018-A01946-49 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2020-05-28; First posted 2020-11-20 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Bariatric Surgery; Long Term Follow-Up; Weight Regain
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Multi-centre, randomised, open, controlled study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Active Comparator): In the control group, patients will follow a care pathway respecting the current recommendations : a systematic clinical visit scheduled each year with the multidisciplinary team.
  Interventions: Other: Control Group
- Experimental Group (Experimental): In the intervention group, patients will follow a new care pathway with visits triggered by weight evolution
  Interventions: Other: Intervention Group

INTERVENTIONS:
Other: Control Group — Clinical visits conducted by a multidisciplinary team every year
  Other Names: Clinical visits conducted by a multidisciplinary team every year
  Arms: Control Group
Other: Intervention Group — Clinical visits are triggered by weight evolution measured by connected balance
  Other Names: Clinical visits triggered by weight evolution
  Arms: Experimental Group

SUMMARY:
Current guideline recommend yearly multidisciplinary postoperative follow-up after bariatric surgery. However, practices remain very heterogeneous, and only a fraction of patients are still follow-up beyond two years after the operation.

This study will assess a new care pathway in which the patients are follow-up according to the weight evolution measured by the patient using a connected scale.

DETAILED DESCRIPTION:
Bariatric surgery is developing rapidly. In France, the number of annual interventions increased threefold between 2001 and 2015, from 16,000 to 50,000 per year. This rapid development is explained by the well-demonstrated benefits of surgery: spectacular improvement in the quality of life, reduction in co-morbidities (diabetes, cardiovascular diseases, and steatohepatitis), and significant reduction in mortality linked to severe obesity. However, the benefits of surgery may decrease over time and may be associated with side effects.

Current guideline recommend yearly multidisciplinary postoperative follow-up after bariatric surgery. However, practices remain very heterogeneous, and only a fraction of patients are still follow-up beyond two years after the operation. The current recommendations therefore do not seem adapted to clinical reality. They do not prevent the regain of weight in many patients, which frequently leads to re-operations. Even more worrying is the possible occurrence of late complications, sometimes serious and life-threatening.

This study will assess a new care pathway in which the patients are follow-up according to weight evolution measured by the patient using a connected scale.

ELIGIBILITY:
Inclusion Criteria:

Patients aged> = at 18 years old Patients who have benefited from a Roux-en-Y Gastric By-Pass or Sleeve Gastrectomy bariatric surgery 2 years ago Preoperative Body Mass Index between 35 kg/m2 and 59 kg/m2 Access to the wired network at home. Social insured patient Patient who signed the informed consent

Exclusion Criteria:

Lack of autonomy for the use of remote monitoring equipment or psychological or psychiatric disorders making it difficult to optimally use the remote monitoring equipment

Administrative reasons: inability to receive informed consent information, inability to participate in the entire study, lack of social security coverage, refusal to sign consent, patient under guardianship or justice system.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 390 (Estimated)
Dates: Start 2021-03-25 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Evaluate the efficacy of new care pathway | 3 years
  The main evaluation criterion is the success rate in terms of weight loss defined by an excess weight loss greater than 50%, in the absence undernutrition.
  Undernutrition is defined by a BMI < 21 kg / m2 and / or an albumin level <35 g /l

SECONDARY OUTCOMES:
Cost-effectiveness of new care pathway | 3 years
  Cost-effectiveness of new care pathway
Number of visits made by the multidisciplinary team | 3 years
  Number of visits made by the multidisciplinary team
Number of postoperative surgical and / or medical complications | 3 years
  Number of postoperative surgical and / or medical complications that justified hospitalisation
Change of nutritional parameters in the blood of vitamines | 3 years
Change of nutritional parameters in the blood of minerals | 3 years
Change of nutritional parameters in the blood of protein | 3 years
Dutch Eating Behavior Questionnaire (DEBQ) | 3 years
  Dutch Eating Behaviour Questionnaire (DEBQ) consists of 33 items and assesses on a 5-point Likert scale, ranging from "never" to "very often" external, restraint and emotional eating. For the study, only the 10 items of the external eating subscale will be used. The variable of interest will be the corresponding External eating subscale score.
Frequency of Food Consumption Questionnaire | 3 years
  A food frequency questionnaire (FFQ) consists of a finite list of foods and beverages with response categories to indicate usual frequency of consumption over the time period queried. To assess the total diet, the number of foods and beverages queried typically ranges from 80 to 120.
Anxiety and depression by Hospital Anxiety and Depression Scale questionnaire (HAD) | 3 years
  Changes of anxiety and depression over three weeks training on a 4-point likert scale scored 0-3. Max 21 Points for each subscale, cut off for anxiety and Depression are set at 7 Points higher values represent more anxiety and Depression.
Ricci-Gagnon score | 3 years
  Evaluation of physical activity This score describe the physical profile : inactive, active, very active, at month 4 It is calculated by adding the number of points (1 to 5) corresponding to the box checked for each question.
  Less than 18=inactive Between 18 and 35=active More than 35=Active
Quality of life of SF36 | 3 years
  Short Form 36 v2.0 acute (SF-36) is a 36-item, patient-reported survey of patient health. SF-36 measures the subject's overall Health Related Quality of Life on 8 domains: physical functioning, role functioning, bodily pain, general health, vitality, social functioning, role emotional and mental health.
Quality of life of questionnaire EQ-5D-5L | 3 years
  The EQ-5D-5L questionnaire will be used to estimate the impact on subjects' health-related quality of life and provides a description of subjects' problems by dimensions (descriptive system), a score for overall self-rated health (visual analogue scale [VAS]) as well as an index score (EQ-5D-5L index). EQ-5D index score range: 0 to 1 and EQ-5D-VAS: range 0 to 100. A higher score indicates better self reported health status.

CONTACTS AND LOCATIONS:
Overall Officials: François Pattou, MD,PhD, Principal Investigator — University Hospital, Lille
Locations (2):
- France (2):
  - Ch Boulogne-Sur-Mer - Boulogne Sur Mer, Boulogne-sur-Mer
  - Hop Claude Huriez Chu Lille, Lille